CLINICAL TRIAL: NCT03672136
Title: Concurrent Chemoradiotherapy Combination With Anlotinib for Unresectable Stage III NSCLC Patients：An Exploratory Single-Arm Phase II Clinical Trail
Brief Title: Concurrent Chemoradiotherapy Combination With Anlotinib for Unresectable Stage III NSCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Chief Physician, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER0300
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent Chemoradiotherapy+Anlotinib (Experimental): 1. Radiotherapy: Thoracic radiotherapy dose will be 2.0Gy per day, given 5 days a week, to cumulative dose of 60～66Gy. If radiotherapy and chemotherapy are conducted in the same day, chemotherapy should be priority to radiotherapy.
  2. Chemotherapy: Platinum based dual drug regime determined by researcher.After finishing concurrent chemoradiotherapy, there is no need of maintenance chemotherapy.
  3. Anlotinib: Combined with 12mg/d QD Anlotinib on the first, second weeks and fourth, fifth weeks of radiotherapy, that is on the day1~14, day22~36.
  4. Maintenance therapy: One month after finishing concurrent chemoradiotherapy, 12mg/d QD Anlotinib can be administrated, each cycle is defined as 2 weeks on-treatment followed by 1 week off-treatment. The treatment can continue until disease progression or treatment intolerance, but should not exceed 24 months.
  5. During the course of study, it's not allowed to receive other anti-tumor therapy.
  Interventions: Drug: Anlotinib; Other: Concurrent Chemoradiotherapy

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a novel multi-target tyrosine Kinase inhibitor that inhibits VEGFR2/3, FGFR1-4, PDGFD α/β, c-Kit and Ret.
Other: Concurrent Chemoradiotherapy — Concurrent chemoradiotherapy as the current standard of care for unresectable stage III non small cell lung cancer patients

SUMMARY:
The purpose of this study is to determine whether concurrent chemoradiotherapy combination with Anlotinib is safe, effective in the treatment of unresectable stage III NSCLC patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether concurrent chemoradiotherapy combination with Anlotinib is safe, effective in the treatment of unresectable stage III NSCLC patients, whether this regimen can improve PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, signed informed consent.
2. Patients pathologically diagnosed as locally advanced (IIIB / IV) unresectable non-small cell lung cancer, with measurable lesions; IIIa3 patient: Multiple stations lymph node metastasis detected by mediastinoscope, other lymph node biopsy or PET-CT; IIIa4 patient: Bulky or stable multiple stations N2 lymph node metastasis (Bulky lymph node: short diameter > 2cm in spiral CT imaging, especially the extranodal invasion); and IIIb patient; T3/4 patient with several ipsilateral or contralateral satellite nodules metastasis will be excluded.
3. Detection of genotypes by providing detectable specimens (tissue) prior to enrollment: patients with negative EGFR mutation, or ALK rearrangement test results.
4. Patients aged between 18 -75 years; with ECOG PS Scoring: 0~1 point; with expected survival time>3 months.
5. Patients with normal organ function within 7 days prior to treatment, the following criteria are met:

   a) blood routine examination criteria (without blood transfusion in 14 days) : i) hemoglobin (HB) ≥100g/L; ii) white blood cell (WBC)≥ 3.0×10e9/L, absolute neutrophil count (ANC) ≥1.5×10e9/L; iii) platelet (PLT) ≥100×10e9/L; b) biochemical tests meet the following criteria: i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr) ≥60mL/min;
6. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥50% lower limit of normal (LLN);
7. Lung function evaluation: forced expiratory volume in first second (FEVI)≥1.45L/s.

Exclusion Criteria(Patient meet any criteria as following will be excluded):

1. Patients who had previously used anlotinib hydrochloride capsules;
2. Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer);
3. Patients with empty lung squamous cell carcinoma, or non-small cell lung cancer with hemoptysis (>20 mL/day);
4. Patients had other malignancies in the past 5 years or currently, except undergone resection and at least 5 years of progression free survival or cured cervical cancer in situ, basal cell carcinoma and superficial bladder tumor;
5. Patients who planned to receive systemic anti-tumor therapy within 4 weeks prior to allocation or during the course of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy, except the immunoregulation agents, such as thymosin and lentinan;
6. Patients with more than common terminology criteria for adverse events (CTC AE) level 1 unmitigated toxicity due to any previous treatment, not including hair loss;
7. Patients have a variety of factors that affect oral medication (such as cannot swallow, chronic diarrhea and intestinal obstruction, etc.);
8. Patients with pleural effusion or ascites, causing respiratory syndrome (≥ CTC AE level 2 dyspnea);
9. Patients with any severe and/or uncontrolled disease, including:

   1. blood pressure control is not ideal (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg);
   2. myocardial ischemic or myocardial infarction, arrhythmia (including QTc ≥480 ms) and ≥ 2 levels of congestive heart failure (NYHA classification);
   3. active or uncontrollable serious infection (≥CTC AE Level 2 infection);
   4. liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need to be treated with antiretroviral therapy;
   5. renal failure requires hemodialysis or peritoneal dialysis;
   6. history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation;
   7. poor control of diabetes (fasting blood glucose [FBG]> 10 mmol/L);
   8. urine routine test protein≥++, and confirmed 24 hours urine protein>1.0 g;
   9. patients with a seizure and need treatment;
   10. Patients with gastric ulcer;
10. Received a major surgical treatment within 28 days prior to allocation, with a biopsy or a significant traumatic injury;
11. Imaging shows that the tumor has been violated around important vascular or the researchers determine the tumor is likely to invade important blood vessels caused by fatal bleeding during the follow-up;
12. Regardless of the severity, patients with any signs or medical history of bleeding; within 4 weeks prior to allocation, patients with any bleeding events ≥ CTC AE level 3, unhealed wounds, ulcers or fractures;
13. Patients with artery/venous thrombotic occurred within 6 months before allocation, such as cerebrovascular accident (including temporary ischemic attack),deep vein thrombosis and pulmonary embolism;
14. Patients with a history of psychotropic medicine abuse and cannot quit or have mental disorders;
15. Patients during pregnancy or lactation period;
16. Patients participated in other anti-tumor drug clinical trials within 4 weeks;
17. According to the determination of researchers, patients were diagnosed with disease which will severely endanger the security of patients or influence the completion of this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression Free Survival

SECONDARY OUTCOMES:
OS | 2 years
  Overall survival
ORR | 2 years
  Objective Response Rate
DCR | 2 years
  Disease Control Rate

CONTACTS AND LOCATIONS:
Overall Officials: JINMING YU, doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- SHANDONG Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pritchard RS, Anthony SP. Chemotherapy plus radiotherapy compared with radiotherapy alone in the treatment of locally advanced, unresectable, non-small-cell lung cancer. A meta-analysis. Ann Intern Med. 1996 Nov 1;125(9):723-9. doi: 10.7326/0003-4819-125-9-199611010-00003. PMID 8929005
- [Result] Bao Y, Peng F, Zhou QC, Yu ZH, Li JC, Cheng ZB, Chen L, Hu X, Chen YY, Wang J, Wang Y, Ma HL, Xu ZM, Lu RB, Deng XW, Chen M. Phase II trial of recombinant human endostatin in combination with concurrent chemoradiotherapy in patients with stage III non-small-cell lung cancer. Radiother Oncol. 2015 Feb;114(2):161-6. doi: 10.1016/j.radonc.2014.11.039. Epub 2014 Dec 9. PMID 25497558
- [Result] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152